CLINICAL TRIAL: NCT03820167
Title: Mitochondrial DNA in Fresh Versus Frozen Embryo Culture Media of Polycystic Ovarian Syndrome Patients Undergoing In Vitro Fertilization
Brief Title: Mitochondrial DNA in Fresh Versus Frozen Embryo Culture Media of PCOS Women Undergoing In Vitro Fertilization
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Principal investigator, Cairo University
Other Study IDs: 49
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Polycystic Ovary Syndrome; Assisted Reproduction
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — embryo culture media from day 3 morphologically good embryos will be collected after embryo transfer of fresh and thawed cycles. The media will be immediately frozen into sterile, PCR clean (free from DNA, DNase, RNase and PCR inhibitors) tubes and stored at - 20 C until nucleic acid purification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fresh sample: Morphologically good embryos will be cultured in a culture dish and the supernatants will be collected freshly from culture system at day 3 and stored at -20 ̊ c until being tested.
  Quantification of mtDNA in fresh and frozen culture media using qPCR technique.
- Frozen embryos: Morphologically good embryos scheduled for freezing will be cryopreserved for less than one year and thawed, the supernatant will be collected and stored at -20 ̊ c until being tested. Quantification of mtDNA in fresh and frozen culture media using qPCR technique.

SUMMARY:
Ninety women with PCOS candidate for ICSI were randomized to 2 groups:Group A: fresh samples of PCOS patients undergoing IVF (no= 45) and Group B: frozen samples of PCOS patients undergoing IVF (no= 45). Morphologically good embryos will be cultured in a culture dish and the supernatants will be collected freshly from culture system at day 3 and stored at -20 ̊ c until being tested. Morphologically good embryos scheduled for freezing will be cryopreserved for less than one year and thawed, the supernatant will be collected and stored at -20 ̊ c until being tested. Quantification of mtDNA in fresh and frozen culture media using qPCR technique.The template DNA prepared and the dilution standards prepared will be used for qPCR to determine the amount of MtDNA and nuclear DNA in the sample using QuantiTect SYBR Green PCR Kit

DETAILED DESCRIPTION:
Ninety women with PCOS candidate for ICSI were randomized to 2 groups:Group A: fresh samples of PCOS patients undergoing IVF (no= 45) and Group B: frozen samples of PCOS patients undergoing IVF (no= 45). Morphologically good embryos will be cultured in a culture dish and the supernatants will be collected freshly from culture system at day 3 and stored at -20 ̊ c until being tested. Morphologically good embryos scheduled for freezing will be cryopreserved for less than one year and thawed, the supernatant will be collected and stored at -20 ̊ c until being tested. Quantification of mtDNA in fresh and frozen culture media using qPCR technique.The template DNA prepared and the dilution standards prepared will be used for qPCR to determine the amount of MtDNA and nuclear DNA in the sample using QuantiTect SYBR Green PCR Kit (Qiagen)

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-35 yrs.
2. BMI: ≤25.
3. PCO: diagnosed by Rotterdam criteria (at least two of the following):

   1. Polycystic ovary morphology with one ovary being sufficient for diagnosis.
   2. Hyperandrogenism: clinically or biochemically.
   3. Anovulation or oligo-ovulation.
4. Gravidity and parity: Nulligravida.
5. Compliance: primary infertility

Exclusion Criteria:

* Known medical problems as diabetes mellitus, hypertension, cardiac, hepatic or renal problem.
* Special habits of medical importance as smoking.
* Other endocrinopathies

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Detailed history taking with special emphasis on:
  1. Personal history (name, age, marital state, parity, address).
  2. Menstrual history (duration, cycle, amount, regularity, last menstrual period).
  3. Medical history for acne and hirsutism.
  Clinical examination with special emphasis on:
  1. Height and weight of the patients to calculate the BMI (weight in kg/ height in m2).
  2. Examinationfor presence of acne and/ or hirsutism (patients with score > 8 on Ferryman & Gallawey score were considered as hirsute).
  3. Ultrasound examination to confirm diagnosis of PCOS (Using the vaginal probe).
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 4 weeks after embryo transfer
  detection of intrauterine gestational sac by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Ganna IVF center, Giza, Cairo Governorate, Egypt